CLINICAL TRIAL: NCT06059144
Title: Induced Hypertension in Acute PRogrESsive Perforating Artery Stroke Using Peripheral Dilute noREpinephrine
Acronym: PRESSURE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2022/23
Record Dates: First submitted 2023-05-26; First posted 2023-09-28 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Acute; Stroke, Ischemic
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induced hypertension using norepinephrine (Experimental): Standard care and peripheral intravenous norepinephrine. Norepinephrine (dilution: 10µg/ml, initial dose: 0.04µg/kg/min) will be titrated until MAP is between 110 and 120mmHG (with a maximal systolic blood pressure of 210mmHG) Gradually decrease of norepinephrine will start after 24h of NIHSS stabilization.
  Standard care includes antithrombotic treatments according to the physician's choice and ESO recommendations
  Interventions: Drug: Peripheral intravenous norepinephrine
- Standard care (No Intervention): Standard care includes antithrombotic treatments according to the physician's choice and ESO recommendations

INTERVENTIONS:
Drug: Peripheral intravenous norepinephrine — Norepinephrine (dilution: 10µg/ml, initial dose: 0.04µg/kg/min) will be titrated until MAP is between 110 and 120mmHG (with a maximal systolic blood pressure of 210mmHG) Gradually decrease of norepinephrine will start after 24h of NIHSS stabilization.
  Arms: Induced hypertension using norepinephrine

SUMMARY:
PRESSURE is a multicenter, prospective, randomized, open, blinded end-point assessed (PROBE) trial, that aims to evaluate the efficacy and safety of drug-induced hypertension using peripheral dilute norepinephrine, in patients with acute ischemic stroke in a perforating artery territory and experiencing early neurological deterioration.

DETAILED DESCRIPTION:
Perforating artery strokes represent 25% of all ischemic strokes and is a well-known cause of progressive symptoms : 12 to 36% of cases experience early neurological deterioration in hours or days after stroke onset. A possible mechanism is hypoperfusion due to lack of a rapid development of collateral flow because of the terminal distribution of perforating arteries. Moreover, arterioles are maximally dilated within penumbra region, resulting in a cerebral autoregulation failure and a passive dependence of cerebral blood flow on arterial pressure. Thus, induced-hypertension therapy by using vasopressive agents is an attractive therapy to increase the cerebral perfusion pressure and therefore restore blood flow in the ischemic penumbra.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke < 72 h in a perforating artery territory on brain MRI
* Early neurological deterioration or fluctuation, attested by the neurologist in charge, defined by a ≥ 3-point increase in global NIHSS score OR a 2-point increase on motor or ataxia score, whether this deterioration is transient or permanent.
* Time between early neurological deterioration and randomization < 6 hours
* Age ≥ 18 years
* Contraception required in women of childbearing potential (Intra-uterine device, hormonal contraception associated with inhibition of ovulation (combined or progestogen-only; oral, intravaginal or transdermal), Female Sterilization, Vasectomised partner, sexual abstinence)
* Beneficiary of a health insurance system

Exclusion Criteria:

* - Pre-Stroke Modified Rankin Score > 3
* Contraindication to brain Magnetic Resonance Imaging (MRI)
* High risk of intracerebral hemorrhage:

  * Cerebral microbleeds ≥ 10
  * Non traumatic focal superficial siderosis
  * Hemorrhagic transformation of the present ischemic stroke
  * Previous history of intracerebral hemorrhage (symptomatic or asymptomatic identified on brain MRI)
  * Intracranial vascular malformation or tumor with suspected risk of rupture or bleeding
* Prior intravenous thrombolysis < 24 hours
* Requirement for anticoagulation in the first 7 days after randomization
* Systolic blood pressure (SBP) > 180mmHG and/or mean arterial pressure (MAP) ≥ 110mmHG at inclusion
* Large artery atherosclerosis (ipsilateral atherosclerotic stenosis > 50%), intra and extracranial dissection, or cardio-embolic stroke mechanisms
* Drugs with important interactions with norepinephrine: monoamine oxidase inhibitors (including reversible, non-selective agents such as linezolid), tricyclic antidepressants, entacapone.
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-08-28 (Estimated); Study Completion 2027-11-28 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) | Day 0
  Functional independence defined by modified Rankin scale 0-2 or return to pre-stroke modified Rankin scale, assessed at 90 days. The assessment of the clinical outcome at 90 (±15) days will be conducted by an independent qualified assessor (blinded to patient treatment allocation). The minimal value of the modified Rankin Scale is 0 (best outcome) and the maximum value is 6 (worst outcome).
modified Rankin Scale (mRS) | Day 90
  Functional independence defined by modified Rankin scale 0-2 or return to pre-stroke modified Rankin scale, assessed at 90 days. The assessment of the clinical outcome at 90 (±15) days will be conducted by an independent qualified assessor (blinded to patient treatment allocation). The minimal value of the modified Rankin Scale is 0 (best outcome) and the maximum value is 6 (worst outcome).

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) | Day 90
  Functional outcomes as measured through the ordinal (shift) modified Rankin scale. The minimal value of the modified Rankin Scale is 0 (best outcome) and the maximum value is 6 (worst outcome).
modified Rankin Scale (mRS) | Day 90
  Functional outcomes as measured through the rate of 90-day excellent functional outcome (mRS 0-1). The minimal value of the modified Rankin Scale is 0 (best outcome) and the maximum value is 6 (worst outcome).
NIHSS Score | Day 0
  c. Early neurological improvement defined as a reduction (compared to the NIHSS at the time of randomization) of at least 3 points or a score of 0 or 1 on the NIHSS
NIHSS Score | Day 7
  Early neurological improvement defined as a reduction (compared to the NIHSS at the time of randomization) of at least 3 points or a score of 0 or 1 on the NIHSS
Mortality | Day 90
Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) | Day 90
  The minimum value of the PC-PTSD-5 is 0 (best outcome) and the maximum value is 5 (worst outcome)
Hospital Anxiety and Depression Scale | Day 90
  The HAD scale provides 2 sub-scores, one on depression, and one on anxiety. Both sub-scores range from 0 (best outcome) to 21 (worst outcome)
Proportion of patients presenting Acute coronary syndrome | Day 7
  Acute Coronary Syndrome refers to ST elevation myocardial infarction (STEMI), non-ST elevation myocardial infarction (NSTEMI), and unstable angina. We will estimate the proportion of patients presenting at least one of these events until day 7.
Proportion of patients presenting Congestive heart failure | Day 7
  We will estimate the proportion of patients presenting at least one episode of congestive heart failure until day 7.
Proportion of patients presenting Tachyarrhythmia | Day 7
  Tachyarrythmia refers to a resting heart rate that exceeds 100 beats per minute. We will estimate the proportion of patients presenting at least one episode of tachyarrythmia until day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline RENOU, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided